CLINICAL TRIAL: NCT06272942
Title: Identifying Post ICU Morbidity in Patients With ARDS in the United States
Brief Title: An Observational Study to Identify New Health Problems Arising After an Intensive Care Unit Admission in People With Acute Respiratory Distress Syndrome in the United States
Acronym: SeeMe Tool
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22722
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Post Intensive Care Syndrome (PICS)
MeSH Terms: conditions — Respiratory Distress Syndrome; postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Post intensive care unit (ICU) morbidity: All adult patients in Optum Claims data from January 1, 2016 until October 1, 2022.
  Interventions: Other: An ICU admission and a temporally related ARDS diagnosis

INTERVENTIONS:
Other: An ICU admission and a temporally related ARDS diagnosis — This is a disease study to learn more about the morbidity after an ICU admission and a temporally related ARDS diagnosis.
  ARDS stands for acute respiratory distress syndrome.

SUMMARY:
This is an observational study in which data already collected from people with acute respiratory distress syndrome (ARDS) admitted to an intensive care unit (ICU) are studied.

ARDS is a life-threatening condition in which fluid builds up in the lungs making breathing difficult.

In observational studies, only observations are made without participants receiving any advice or any changes to health care.

People who are admitted to ICU for serious illnesses, like ARDS, often experience new health problems during and after their ICU stays. These health problems that may include physical, mental, and/or emotional disorders, are called post-intensive care syndrome (PICS). Identifying these new health problems early can help people by timely treatments and care.

In this study, researchers want to identify any health problems that arise after ICU admission in people with ARDS in the United States (US). To do this, researchers will collect information on health problems, treatments, medicines, and healthcare visits in people with ARDS, 1 year before and after an ICU admission.

They will then look to see whether the health problems are in areas that have been described as the post intensive care syndrome (PICS).

In addition, they will measure healthcare related costs in the one year after admission and compare it to the one year prior to admission.

Researchers will also compare this information with data collected for people with pneumonia who did not require ICU admission. This will help them to identify any new health problems arising due to ICU stays.

The data will come from participants' medical claims information stored in the Optum Clinformatics Data Mart database from 2016 to 2022. The claims data will only be collected for people in the US.

Researchers will collect data from participants admitted to ICU for ARDS for a maximum of 1 year before and after their stay.

ELIGIBILITY:
Inclusion Criteria:

* continuous coverage of at least 365 days (>= 1 year) pre-index date for the cohort
* age >= 18 years
* not seen outside the healthcare system

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients in Optum Claims data with acute respiratory distress syndrome (ARDS) admitted to an intensive care unit (ICU) from January 1, 2016 until October 1, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 140000 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Morbidity | at 1,3,6 and 12 month pre- and post- index hospital admission
  Morbidity will be stratified by comorbidities, procedures, medications, healthcare utilization.
Post ICU Syndrome-related morbidity | at 12 months post- index hospital admission
  PICS-related morbidity will be stratified by comorbidities, procedures, medications, healthcare utilization.
  PICS stands for post intensive care unit syndrome.
Incident morbidity | at 1, 3, 6 and 12 months post- index hospital admission
  Incident morbidity will be stratified by comorbidities, procedures, medications, healthcare utilization.
Post ICU Syndrome-related incident morbidity | at 1, 3, 6 and 12 months post- index hospital admission
  PICS-related incident morbidity will be stratified by comorbidities, procedures, medications, healthcare utilization.
Difference in prevalence rates pre versus post index hospitalization | at 1, 3, 6 and 12 months post- index hospital admission
Average total healthcare costs based on healthcare billing data in the one year post index ICU admission | at 12 months post- index hospital admission
  Average total healthcare costs will be based on healthcare billing data in the one year post index ICU admission.

OTHER OUTCOMES:
Exploratory, descriptive difference in ranking of PICS domain comorbidity ratios observed for ARDS (ICU admissions) versus pneumonia (non ICU admissions). | At 1, 3, 6 and 12 months post-index admission
  Descriptive analyses will be performed and trajectories of post ARDS (ICU admission) versus pneumonia (non ICU admission) will be compared visually using waterfall plots.
  ARDS stands for acute respiratory distress syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.